CLINICAL TRIAL: NCT01653756
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multi-Dose, Cross-Over, Efficacy and Safety Study of Duvelisib in Mild Asthmatic Subjects Undergoing Allergen Challenge
Brief Title: A Phase 2a, Efficacy and Safety Study of Duvelisib in Mild Asthmatic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IPI-145-03; 2012-001729-28 (EudraCT Number)
Record Dates: First submitted 2012-07-19; First posted 2012-07-31 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: Asthma; Allergen Challenge
MeSH Terms: conditions — Asthma | interventions — duvelisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPI-145 (Active Comparator): Capsules
  Interventions: Drug: IPI-145, a PI3K Inhibitor; Drug: Placebo to match IPI-145
- Placebo (Placebo Comparator): Capsules
  Interventions: Drug: IPI-145, a PI3K Inhibitor; Drug: Placebo to match IPI-145

INTERVENTIONS:
Drug: IPI-145, a PI3K Inhibitor — Active drug
Drug: Placebo to match IPI-145 — Comparator

SUMMARY:
The purpose of this study is to examine the effects of multi-dose regimens of IPI-145 on lung function in mild asthmatic subjects following allergen challenge.

DETAILED DESCRIPTION:
This is a phase 2a, randomized, double-blind, placebo-controlled, multi-dose, 2-way cross-over study designed to examine the effect of IPI-145 on lung function and inflammatory indices in mild, allergen-reactive asthmatic subjects undergoing allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults between 18 and 60 years of age
* Diagnosis of asthma (mild) for at least 6 months prior to Screening
* Forced expiratory volume in one second (FEV1) ≥70% of predicted value at Screening
* A positive skin prick test to test allergen

Exclusion Criteria:

* Any prior treatment with a phosphoinositide-3-kinase (PI3K) inhibitor other than IPI-145 in a previous clinical study
* Acute asthma exacerbations within 6 weeks prior to Screening
* Use of any medication for the treatment of asthma other than a short-acting β2 agonist (as needed) within the 4 weeks prior to Screening
* Participation in another clinical study within minimum of 30 days prior to study Screening
* A positive screen result for active or latent tuberculosis
* A history of cardiovascular disease
* The concomitant use of acid-reducing agents and cholinesterase inhibiting medication
* Inadequate hepatic function defined by Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) greater than 1.5 times greater limit of normal (ULN)
* Inadequate renal function defined by serum creatinine greater than 2.0 milligrams/dL

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1) | Day 14

SECONDARY OUTCOMES:
Maximum concentration (Cmax), Area Under the Curve, and terminal elimination half-life (T1/2) pre-dose and up to 12 hours post dose | Day 14
Number of Participants with Adverse Events as a Measure of Safety | From signing of informed consent through 21 days following study drug administration
Change in C-reactive Protein (CRP) levels | Screening and/or Day 1 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (4):
- Germany (3):
  - Investigational Site, Berlin
  - Investigational Site, Großhansdorf
  - Investigational Site, Wiesbaden
- Investigational Site, Harrow, United Kingdom